CLINICAL TRIAL: NCT06013683
Title: Mastocvtosis Collaborative Network of China: A Registry for Patients With Systemic Mastocytosis
Brief Title: A Registry for Patients With Systemic Mastocytosis in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Director, Clinical Professor, The First Affiliated Hospital of Soochow University
Other Study IDs: SZ-SM01
Record Dates: First submitted 2023-07-23; First posted 2023-08-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Systemic Mastocytoses
MeSH Terms: conditions — Mastocytosis, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Registry for Patients With Systemic Mastocytosis in China is a voluntary, observational database that will capture demographic, socioeconomic, and disease information with systemic mastocytosis. No experimental intervention is involved.

DETAILED DESCRIPTION:
Systemic Mastocytosis (SM) is an extremely rare and heterogeneous spectrum of diseases characterized by the buildup of genetically altered mast cells in bone marrow sections and/or other extracutaneous organ(s). SM has not been given enough attention in China at present, and the epidemiological data in China are not clear. To understand the epidemiological characteristics and distribution patterns of SM patients in China. To establish a China-wide database platform for registering SM patients and to develop uniform registration standards and processes; to register SM patients who meet the enrollment criteria nationwide through a multicenter collaborative approach and to collect information on their baseline data, clinical manifestations, laboratory tests, treatment regimens, and follow-up results; to perform quality control and data cleansing on the information collected in the registration database, as well as to perform descriptive and inferential statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a diagnosis of systemic mastocytosis according to World Health Organization (WHO) classification, including subtypes of SM, who is willing and able to provide written online informed consent.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of systemic mastocytosis according to World Health Organization (WHO) classification, including subtypes of SM, who is willing and able to provide written online informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The morbidity rate over 2 years ofSystemic Mastocytosis and its subtypes (cases per 1,000 individuals per year) | at 2 year
  Evaluation of the morbidity rate over 2 years of Systemic Mastocytosis and its subtypes including Bone marrow mastocytosis (BMM), Indolent SM, Smoldering SM, Aggressive SM, SM with an associated hematologic neoplasm and Mast cell leukemia. (cases per 1,000 individuals per year)

SECONDARY OUTCOMES:
Demographic characteristics of Systemic Mastocytosis | at 2 year
  1. The median age of Systemic Mastocytosis patients (year-old);
  2. The sex distribution of Systemic Mastocytosis patients (M/F ratio[0-1]);
  3. The ECOG score of Systemic Mastocytosis patients (score[0-5]);
  4. The geographic distribution of Systemic Mastocytosis patients (% per province[0-100]);
Hematological characteristics of Systemic Mastocytosis | at 2 year
  1. The neutrophils, eosinophils, basophils, and mast cells in WBC classification (%);
  2. The proliferative degree in sections of BM (%);
  3. The ratio of mast cells in BM smear and FCM (%);
  4. The ratio of expression of CD25, CD2, and CD30 in FCM (%);
  5. The serum tryptase level(%).
Nonhematological characteristics of Systemic Mastocytosis | at 2 year
  1. The incidence of extramedullary organ infiltration including skin, bone and other organs (%);
  2. The incidence of enlarged liver (%);
  3. The incidence of enlarged spleen (%);
  4. The incidence of enlarged lymphnodes (%);
  5. The incidence of hypoproteinemia and loss weight (%).
Responses to therapy of Systemic Mastocytosis | at 2 year
  1. The rate of eligible complete remission (CR) patients(%);
  2. The rate of eligible partial remission (PR) patients(%);
  3. The rate of eligible clincal improvement (CI) patients(%);
  4. The rate of eligible stable disease (SD) patients(%);
  5. The rate of eligible progressive disease (PD) patients(%);
  6. The rate of eligible loss of reponse (LOR) patients(%).
Survival Distribution of Systemic Mastocytosis | at 2 year
  1. Overall survival (months): Measured the time from enrollment to the date of the last follow-up or death;
  2. Event-free survival (months): Measured the time from the date of attaining CR1 until the first relapse, death, or the final follow-up day.

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, Professor, Principal Investigator — The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China